CLINICAL TRIAL: NCT00540748
Title: Is Oxytocin Given During Surgical Procedure for Abortion Before 12 Weeks of Pregnancy Useful ?
Brief Title: Is Oxytocin Given During Surgical Procedure for Abortion Before 12 Weeks of Pregnancy Useful?
Acronym: oxystudien
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Asker & Baerum Hospital (Other)
Responsible Party: Administrator Marit Kristoffersen, Asker and Baerum Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 392-06154 1.2006.1683 (REK); 392-06154 1.2006.1683 (REK)
Record Dates: First submitted 2007-10-04; First posted 2007-10-08 (Estimated); Last update posted 2010-04-16 (Estimated); Status verified 2009-05

CONDITIONS: Induced Abortion
Keywords: first trimester abortion; oxytocin
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- A1 (Experimental)
  Interventions: Drug: oxytocin
- A2 (No Intervention)

INTERVENTIONS:
Drug: oxytocin — 5 U i.v. during surgical abortion
  Arms: A1

SUMMARY:
This is a randomized, single-blind study using oxytocin 5U i.v. during surgical abortion in one arm of the study, and no medication in the other arm of the study. Comparison is done between the two groups measuring the following outcomes: pain, nausea and blood loss. The investigators' hypothesis is that there will be no significant differences between the two groups.

DETAILED DESCRIPTION:
All women seeking surgical abortion before 12 weeks of pregnancy will be invited to participate in the study. We will include 400 patients. Written consent is given. Pain is measured on a VAS-scale (1-10) 2 hours post operatively and repeated 2 days postoperatively. Nausea is categorized in 4 groups, from 1 (no nausea) to 4 (pronounced nausea with vomiting)and is registered together with bloodloss also during the hospital stay (2 hours) and 2 days postoperatively. The two groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* seeking legal abortion
* first trimester
* surgical intervention
* no current medication
* fluent in norwegian language

Exclusion Criteria:

* current medication
* medical condition with coagulopathy

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2007-10; Primary Completion 2009-06 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
blood loss, pain, nausea | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Annelill Valbo, consultant, MD PhD, Study Director — Kvinneklinikken SABHF
Locations (1):
- Kvinneklinikken SABHF, Baerum, Rud, Norway